CLINICAL TRIAL: NCT00852891
Title: Cardiorespiratory Changes in Patients Being Weaned Off Mechanical Ventilation: a Randomized Crossover Clinical Trial
Brief Title: Cardiorespiratory Changes in Patients Being Weaned Off Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Silvia Regina Rios Vieira, Hospital de Clínicas de Porto Alegre
Other Study IDs: 2004341 UFRGS
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Critical Care; Weaning
Keywords: weaning; echocardiogram; diastolic dysfunction; Mechanical ventilation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study was to analyze changes in cardiac function using Doppler echocardiogram in critical patients during weaning from mechanical ventilation using two different weaning methods (pressure support and T-tube) and to compare a subgroup of patients: success vs. failure in weaning and patients with vs. without heart disease.

DETAILED DESCRIPTION:
Weaning from mechanical ventilation (MV) involves physiological changes that can overload the cardiorespiratory system due to changes in the interaction between patient and ventilator.

This was a randomized crossover clinical trial that included patients in an intensive care unit (ICU) who had been on MV for more than 48 hours and who were considered ready for weaning. Cardiorespiratory variables, oxygenation, electrocardiogram (ECG) and Doppler echocardiogram findings were analyzed at baseline and after 30 minutes in each trial weaning method (PSV and T-tube). Comparisons were made between PSV and T-tube, weaning success and failure and patients with and without heart disease, using ANOVA and Student's t test. The level of significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients hemodynamically stable
* conscious (Glasgow scale ≥ 13)
* with adequate gaseous exchange (O2 saturation ≥ 95%, fraction of inspired oxygen (FiO2) ≤ 40% and positive end-expiratory pressure (PEEP) = 5
* with no acidosis or alkalosis)
* normal electrolyte levels
* presence of respiratory drive
* informed consent was signed by the patients and/or family members

Exclusion Criteria:

* hemodynamic instability
* severe intracranial disease
* barotrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving MV for more than 48 hours, who had been admitted to the Intensive Care Unit (ICU), and who met the criteria for weaning from MV according to the parameters previously defined were selected to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2005-12; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia RR Vieira, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil